CLINICAL TRIAL: NCT00392366
Title: The Clinical Evaluation of the Laser Interstitial Thermal Therapy (LITT ), Under "Real Time" MRI Guidance, for the "Minimal Invasive" Treatment of Liver Metastasis - a Phase IIa Mono-centric Study, Without Direct Benefice to the Patient
Brief Title: Laser Interstitial Thermal Therapy Under "Real Time" MRI Guidance for "Minimal Invasive" Treatment of Liver Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioTex, Inc. (Industry)
Responsible Party: Ashok Gowda, BioTex, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LITT / METASTASE HEPATIQUES
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Carcinoma, Hepatocellular; Liver Neoplasms; Digestive System Neoplasms
Keywords: MRI guided Laser Therapy; Laser Interstitial Thermal Therapy; Magnetic Resonance Thermal Imaging; Liver Metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Digestive System Neoplasms

INTERVENTIONS:
Device: MR-guided Laser Interstitial Thermal Therapy System

SUMMARY:
The purpose of this study is to determine if the, MR guided, laser interstitial thermal therapy (LITT) treatment technique can be safety and efficiently used for the human liver metastasis

DETAILED DESCRIPTION:
This new "minimally invasive" technique has been tested so far, with success, on animal brain and prostate tumors. LITT has also tested with success by other teams for the treatment of liver metastasis.

The main purpose of this study is to determine if the Visualase, MR guided, laser interstitial thermal therapy device can be safely and efficiently used for the treatment of human liver metastasis originating from the colon and rectal primary tumors.

As secondary objectives for this clinical study is to explore the tolerance of the treatment and its contra indications.

The clinical trial will include a statistical sample of 25 patients and will run over a period of 24 months. The inclusion period will be of 12 months and the patients will be followed up during a period of 7 days after the intervention.

The clinical trial will be performed at the Cochin University Hospital of Paris and the patients will be coming from the oncology / surgery departments of the hospital.

The patients recruited for this study are those who developed several liver metastasis and are planned for the a surgical resection for part of the liver (where metastasis are located). Prior to the surgical resection, a LITT procedure will be performed on one of the metastasis. After the surgical resection histological analysis will be elaborated to compare the real necrosis volume created by the LITT procedure to the expected predicted volume.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients with liver metastasis, originating from colon and liver cancer and proved by histological analysis
* Patient that are scheduled for a surgical resection of part of the liver,
* Patient having a liver metastasis, originating from colon and rectal cancer, smaller or equal to 3 cm
* Patients having the liver metastasis at a distance of at least 1 cm or from the hepatic capsule or/and from a vascular structure

Exclusion Criteria:

* Patients younger than 18 years old
* Patients presenting contra indication for MRI studies
* Patient presenting contra indication to liver surgery
* Patients who already had other interstitial treatment on the targeted lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-07; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Accuracy of predicted lesion geometry to histologically measured dimensions

CONTACTS AND LOCATIONS:
Overall Officials: Paul Legmann, M.D., Principal Investigator — Cochin Hosptial, Paris, France
Locations (1):
- Hospital Cochin, Paris, France